CLINICAL TRIAL: NCT01213017
Title: The Effect of Certolizumab Pegol in Combination With Methotrexate on MRI Synovitis and Bone Edema and Patient Reported Outcomes as Measured Using an Automated Visit Manager System in Moderate to Severe Rheumatoid Arthritis Patients
Brief Title: The Effect of Certolizumab Pegol on MRI Synovitis and Bone Edema in Rheumatoid Arthritis Patients
Acronym: PICS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oklahoma Medical Research Foundation (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMRF-UCB-5-16-2010
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Certolizumab pegol; Magnetic Resonance Imaging; Rheumatoid Arthritis; RAPID 3
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Certolizumab pegol (Experimental)
  Interventions: Drug: certolizumab pegol

INTERVENTIONS:
Drug: certolizumab pegol — 400mg at week 0, 2 and 4, followed by 200 mg every two weeks for 52 weeks
  Other Names: Cimzia

SUMMARY:
The purpose of this study is to determine whether Certolizumab pegol can rapidly reduce the inflammatory changes and inhibit erosions on hand and wrist MRI in patients with active moderate to severe rheumatoid arthritis.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of CSP used in combination with MTX in patients with active moderate to severe RA by evaluating change from baseline in synovitis and bone edema MRI scores at week 6.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe RA (DAS > 4.4)
* at least two swollen and tender joints in one of the hand/ wrist
* patients must have failed at least one non-biologic or biologic DMARDs
* currently receiving MTX therapy

Exclusion Criteria:

* concomitant diseases or pathological conditions that could interfere and impact the assessment of the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
the change from baseline in synovitis and bone edema RAMRIS score. | 6 weeks

SECONDARY OUTCOMES:
the change from baseline in RAMRIS erosion score | 16 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Olech, MD, Principal Investigator — Oklahoma Medical Research Foundation; Norman B Gaylis, MD, Principal Investigator — Arthritis and Rheumatic Disease Specialties
Locations (2):
- United States (2):
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available